CLINICAL TRIAL: NCT00237341
Title: Assessing Functionality Changes Associated With Patients Who Were Taking Short Acting Opioids Chronically and Who Initiated Treatment With Duragesic® (Fentanyl Transdermal System) for the Management of Chronic Low Back Pain.
Brief Title: Duragesic® (Fentanyl Transdermal System) Functionality Trial in Chronic Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR002446
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; opioid; fentanyl
MeSH Terms: conditions — Low Back Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: fentanyl

SUMMARY:
The purpose of this study is to assess physical functionality changes over a minimum of 9 weeks in patients with non-malignant chronic low back pain who are taking short-acting opioids (narcotic pain medications) for 4 or more weeks, and who start taking the long-acting opioid fentanyl in the form of a transdermal (skin) patch.

DETAILED DESCRIPTION:
Chronic pain (pain that lasts for more than 3 months) can limit physical functioning and negatively affect a person socially and emotionally. Chronic low back pain (that is not caused by cancer) is a very common condition that affects up to a third of people in the US at any time. The primary objective of the trial is to assess functionality changes over a minimum period of 9 weeks using the Oswestry Disability Index (ODI) - a questionnaire to measure disability - in patients with non-malignant chronic low back pain who are taking short-acting opioids chronically, and who initiate treatment with Duragesic® (transdermal fentanyl). The patch delivers fentanyl in doses of 25, 50, 75, or 100 micrograms per hour. The ODI is comprised of 10 sections; each section consists of 6 response alternatives. The 10 scales assessed by the ODI are Pain Intensity, Personal Care (washing, dressing, etc.), Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, and Traveling. The secondary objective is to assess changes in health-related quality of life (HRQoL) over the treatment period using the Total Pain Experience (TPE) subscale of the Treatment Outcomes in Pain Survey (TOPS), a questionnaire designed to measure HRQoL changes in patients with chronic pain. The TOPS contains 112 items that are scored into 16 scales. These scales include: Pain Symptoms, Lower Body Functional Limitations, Upper Body Functional Limitations, Perceived Family/Social Disability, Objective Family/Social Disability, Objective Work Disability, TPE (a combination of 5 other scales), Life Control, Passive Coping, Solicitous Responses, Work Limitations, Fear Avoidance, Patient Satisfaction with Outcomes, Health Care Satisfaction, Vitality, and Mental Health (the last two from a questionnaire known as the Short Form-36, or SF-36. Fentanyl transdermal system (skin patch) in a dosage prescribed by the clinical investigator according to the usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (not related to cancer) for at least 3 months
* current use of short-acting opioid (narcotic pain medication) for at least 4 weeks
* initiating fentanyl transdermal patch.

Exclusion Criteria:

* Confusion or reduced level of consciousness
* skin disease
* malignancies (cancer)
* currently hospitalized
* treated with a long-acting opioid within the last 2 months
* pregnant or breast-feeding
* abusing drugs or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2002-06; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PriCara, Unit of Ortho-McNeil, Inc. Clinical Trial, Study Director — PriCara, Unit of Ortho-McNeil, Inc.

REFERENCES:
- See also: Assessing functionality changes associated with patients who were taking short acting opioids chronically and who initiated treatment with Duragesic® for the management of chronic low back pain. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1130&filename=CR002446_CSR.pdf